CLINICAL TRIAL: NCT05059782
Title: Efficacy and Safety of Involving Field Radiotherapy in the Oligo-lesions(Metastasis/Recurrent/Refractory) of Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Liu Zi, Professor, Xi'an Jiaotong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCR-04
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Cancer; Neoplasm, Ovarian; Ovarian Neoplasm; Ovary Neoplasms; Neoplasm, Ovary; Neoplasms, Ovary; Ovary Neoplasm; Neoplasms, Ovarian; Ovary Cancer; Cancer, Ovarian Stromal; Cancers, Ovary; Ovary Cancers; Cancer, Ovarian; Cancers, Ovarian; Ovarian Cancers; Cancer of Ovary; Cancer of the Ovary
Keywords: oligo-lessions; metastasis; recurrent; refractory; ovarian cancer; radiotherapy; chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Drug Therapy; Immunotherapy; Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Group A (drug treatment group) : Patients accept paclitaxel + platinum or paclitaxel single drug chemotherapy of which paclitaxel 135-175mg/m2, carboplatin AUC=5, cisplatin 40-60mg/m2. The treatment should be repeated every 3 weeks. Other second-line and third-line chemotherapy regimens (dose is not specified) are also allowed. Targeted, immunological or PARPi drugs can be added based on pathological and genetic test results until disease progression, unacceptable toxicity or informed consent withdrawal. Group B (radiotherapy group): IFRT, IMRT or SBRT is applied. Radiotherapy regimen: Involving field PGTV 60Gy-70Gy, 2-3Gy/f,5 times/week. External irradiation techniques and doses can be selected based on the previous experience of each center, but all patients enrolled within the center need to be consistent. Group C (radiotherapy + drug group) : IFRT is the same as group B;Drug therapy: same as group A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (drug treatment group) (Active Comparator): Group A (drug treatment group) : Chemotherapy drugs ,targeted drugs or Immune checkpoint inhibitors are taken throughout the body or a combination of these drugs according to clinical needs is performed when necessary.
  Interventions: Drug: chemotherapy, targeted therapeutics, immunotherapy
- Group B (radiotherapy group) (Experimental): IFRT, IMRT or SBRT is applied. Irradiation techniques and doses can be selected based on the previous experience of each center, but all patients enrolled within the center need to be consistent.
  Interventions: Radiation: IFRT, IMRT or SBRT
- Group C (radiotherapy + drug group) (Experimental): Drug therapy is the same as group A; IFRT is the same as group B.
  Interventions: Drug: chemotherapy, targeted therapeutics, immunotherapy; Radiation: IFRT, IMRT or SBRT

INTERVENTIONS:
Drug: chemotherapy, targeted therapeutics, immunotherapy — Chemotherapy drugs ,targeted drugs or Immune checkpoint inhibitors are taken throughout the body or a combination of these drugs according to clinical needs is performed when necessary.
  Arms: Group A (drug treatment group); Group C (radiotherapy + drug group)
Radiation: IFRT, IMRT or SBRT — IFRT（involving field radiotherapy） IMRT （ intensity modulated radiation therapy） SBRT （stereotactic body radiation therapy）
  Arms: Group B (radiotherapy group); Group C (radiotherapy + drug group)

SUMMARY:
In this study, The researchers sought to explore the efficacy and safety of involving field radiotherapy in the oligo-metastatic/recurrent/refractory ovarian cancer patients among different groups which include drug therapy alone, radiotherapy alone, and drug therapy plus radiotherapy by inviting clinical multi-center participation.

DETAILED DESCRIPTION:
The recurrent or refractory ovarian cancer tends to recur repeatedly at increasingly short intervals, making treatment more and more difficult.Patients often have limited physical capacity to undergo repeated systematic treatment. Currently, NCCN（ national comprehensive cancer network ）guidelines recommend palliative radiotherapy in patients with local recurrence of ovarian cancer. With the progress of IMRT（ intensity modulated radiation therapy ）, SBRT ( stereotactic body radiation therapy ) and other radiotherapy technologies, better local tumor control rate can also be achieved, while minimizing the damage to surrounding normal tissues. In this study, the patients will be divided into groups according to their wishes: group A (drug therapy alone), group B (radiotherapy alone), and group C (radiotherapy plus drug therapy).The researchers sought to explore the the efficacy and safety of involving field radiotherapy in the oligo-metastatic/recurrent/refractory ovarian cancer patients in different groups after treatment by inviting multiple centers to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Evidence of histological diagnosis of ovarian cancer (including fallopian tube cancer and primary peritoneal cancer)
3. Pathology or imaging suggested recurrence, with measurable lesions, and the number of lesions ≤3;
4. No serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney and immune deficiency
5. Cooperative Oncology Group-Status (ECOG Status) score 0-2;
6. Expected survival ≥3 months;
7. Feasible abdomen and pelvic cavity MRI/CT;
8. Good compliance, signed informed consent voluntarily.

Exclusion Criteria:

1. Previous radiotherapy at the target lesion site;
2. History of active inflammatory bowel disease or severe stomach and duodenal ulcers;
3. Human immunodeficiency virus (HIV) infected persons;
4. active hepatitis b (HBVDNA quantitative test results exceed the lower limit), or HCV infection (HCVRNA quantitative test results exceed the lower limit);
5. suffering from serious underlying diseases, including but not limited to active infections requiring systemic medication:
6. patients with a history of other malignant tumors (except cured basal cell carcinoma of the skin);
7. neurological or mental disorders that affect cognitive ability;
8. Patients whose lesions have been evaluated by the investigator and cannot be treated with external irradiation or endovascular radiation therapy;
9. those who cannot follow up regularly as prescribed by the doctor;
10. Other reasons not suitable for participating in this study as judged by the researcher.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Local Control ( LC ) | 6 months
  LC will be measured from the start date of treatment until the date of progressive of the target lesion

SECONDARY OUTCOMES:
Progression-free Survival ( PFS ) | 24 months
  PFS is defined as the time from first day of treatment until the first date of either objective disease progression or death due to any cause
Overall Survival ( OS ） | 24 months
  OS is defined as the time from first day of treatment until the date of death due to any cause or the deadline for the study
Rate of Radiation-related Adverse Reactions | 24 months
  Rate of acute and late adverse reactions associated with radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zi Liu, Ph.d, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China